CLINICAL TRIAL: NCT07013487
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Immunogenicity, and Efficacy of V181 Dengue Vaccine in Healthy Participants 2 to 17 Years of Age
Brief Title: A Study to Evaluate V181 Dengue Vaccine in Healthy Participants 2 to 17 Years of Age (V181-005/MOBILIZE-1)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V181-005; MOBILIZE-1 (Other: MSD); 2022-003483-25 (EudraCT Number)
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V181 (Experimental): Participants will receive a single 0.5 mL subcutaneous (SC) dose of V181 on Day 1.
  Interventions: Biological: V181
- Placebo (Placebo Comparator): Participants will receive a single 0.5 mL SC dose of placebo on Day 1.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: V181 — Participants will receive a single 0.5 mL SC dose of V181 on Day 1.
  Arms: V181
Biological: Placebo — Participants will receive a single 0.5 mL SC dose of placebo on Day 1.
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate that V181 is safe and well tolerated, elicits an immune response, and reduces the frequency of virologically confirmed dengue (VCD) of any severity, due to any of the 4 dengue serotypes, regardless of dengue serostatus at baseline in children 2 to 17 years of age.

DETAILED DESCRIPTION:
The Reactogenicity and Immunogenicity Subset consists of approximately 3600 participants who will be followed for immunogenicity and safety through 28 days postvaccination. The Long-term Immunogenicity Subset consists of approximately 620 participants randomly selected from the Reactogenicity and Immunogenicity Subset and will evaluate virus reduction neutralization test (VRNT) at designated timepoints up to 5 years postvaccination.

ELIGIBILITY:
The key Inclusion Criteria include but are not limited to:

* Is generally healthy based on medical history and physical examination.

The key Exclusion Criteria include but are not limited to:

* Has a known or suspected impairment of immunological function.
* Has a history of congenital or acquired immunodeficiency.
* Has a documented human immunodeficiency virus (HIV) infection or is breastfeeding from a mother with documented HIV infection.
* Has a documented history of hepatitis B or C infection.
* Has a bleeding disorder contraindicating subcutaneous vaccination or repeated venipuncture.
* Has a serious or progressive disease, including but not limited to cancer, uncontrolled diabetes, severe cardiac, renal or hepatic insufficiency, or systemic autoimmune or neurologic disorders.
* Has a known neurologic or cognitive behavioral disorder, including encephalitis/myelitis, acute disseminating encephalomyelitis, pervasive development disorder, and related disorders.
* Previous receipt of a dengue vaccine or plans to receive any dengue vaccine (investigational or approved) for the duration of the study (other than the study vaccine).
* Is expected to require systemic corticosteroids ≤28 days after receipt of study intervention.
* Has received a blood transfusion or blood products, including immunoglobulins, ≤6 months before receipt of study intervention or plans to receive a blood transfusion or blood products (including immunoglobulins) ≤28 days after receipt of study intervention.
* Has received immunosuppressive therapies, including chemotherapeutic agents used to treat cancer or other conditions, treatments associated with organ or bone marrow transplantation, or autoimmune disease, ≤6 months before receipt of study intervention or plans to receive immunosuppressive therapies ≤28 days after receipt of study intervention.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12000 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2032-02-02 (Estimated); Study Completion 2032-02-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing a Medically Attended Adverse Event (MAAE) | Up to approximately 6 months postvaccination
  A MAAE is an adverse event (AE) in which medical attention is received during an unscheduled, non-routine outpatient visit, such as an ER visit, office visit, or an urgent care visit with any medical personnel for any reason.
Percentage of Participants Experiencing a Serious Adverse Event (SAE) | Up to approximately 5 years postvaccination
  An SAE is an AE that results in death, is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment.
Reactogenicity and Immunogenicity Subset: Percentage of Participants Experiencing Solicited Injection-site AEs | Up to approximately 5 days postvaccination
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study treatment. Solicited injection-site AEs will include pain/tenderness, erythema/redness, and swelling.
Reactogenicity and Immunogenicity Subset: Percentage of Participants Experiencing Solicited Systemic AEs | Up to approximately 28 days postvaccination
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study treatment. Solicited systemic AEs will include rash, headache, tiredness (fatigue), muscle aches all over body (myalgia), joint pain and fever (pyrexia).
Percentage of Participants Experiencing Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD of Any Severity, Due to Any of the 4 Dengue Serotypes, Regardless of Dengue Serostatus at Baseline | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by wild type (WT) reverse transcription polymerase chain reaction (RT-PCR) or non-structural protein 1 (NS1) enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Percentage of Participants Experiencing Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD of Any Severity, Due to Each of the 4 Dengue Serotypes, Regardless of Dengue Serostatus at Baseline | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD of Any Severity, by Dengue Serostatus at Baseline, Up to Approximately 3 Years Postvaccination | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD of Any Severity, by Dengue Serostatus at Baseline, Up to Approximately 5 Years Postvaccination | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD of Any Severity, Regardless of Dengue Serostatus at Baseline | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD Meeting Criteria for Warning Signs or Severe Dengue, Regardless of Dengue Serostatus at Baseline, Up to Approximately 3 Years Postvaccination | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA. Clinical evaluation for presence of dengue with warning signs or severe dengue will be conducted by an investigator or medically qualified designee, based on pre-specified criteria.
Percentage of Participants Experiencing Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD Meeting Criteria for Warning Signs or Severe Dengue, by Dengue Serostatus at Baseline, Up to Approximately 3 Years Postvaccination | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA. Clinical evaluation for presence of dengue with warning signs or severe dengue will be conducted by an investigator or medically qualified designee, based on pre-specified criteria.
Percentage of Participants Experiencing Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD Meeting Criteria for Warning Signs or Severe Dengue, Regardless of Dengue Serostatus at Baseline, Up to Approximately 5 Years Postvaccination | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA. Clinical evaluation for presence of dengue with warning signs or severe dengue will be conducted by an investigator or medically qualified designee, based on pre-specified criteria.
Percentage of Participants Experiencing Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD Meeting Criteria for Warning Signs or Severe Dengue, by Dengue Serostatus at Baseline, Up to Approximately 5 Years Postvaccination | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA. Clinical evaluation for presence of dengue with warning signs or severe dengue will be conducted by an investigator or medically qualified designee, based on pre-specified criteria.
Percentage of Participants Experiencing Hospitalization Resulting from Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD of Any Severity, Regardless of Dengue Serostatus at Baseline, Up to Approximately 3 Years Postvaccination | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Hospitalization Resulting from Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD of Any Severity, by Dengue Serostatus at Baseline, Up to Approximately 3 Years Postvaccination | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Hospitalization Resulting from Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD of Any Severity, Regardless of Dengue Serostatus at Baseline, Up to Approximately 5 Years Postvaccination | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Hospitalization Resulting from Symptomatic (Requiring Fever on at Least 2 of 3 Consecutive Days) VCD of Any Severity, by Dengue Serostatus at Baseline, Up to Approximately 5 Years Postvaccination | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Symptomatic (Regardless of Fever) VCD of Any Severity, Regardless of Dengue Serostatus at Baseline, Up to Approximately 3 Years Postvaccination | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Symptomatic (Regardless of Fever) VCD of Any Severity, by Dengue Serostatus at Baseline, Up to Approximately 3 Years Postvaccination | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Symptomatic (Regardless of Fever) VCD of Any Severity, Regardless of Dengue Serostatus at Baseline, Up to Approximately 5 Years Postvaccination | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Symptomatic (Regardless of Fever) VCD of Any Severity, by Dengue Serostatus at Baseline, Up to Approximately 5 Years Postvaccination | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Symptomatic (Regardless of Fever) VCD Meeting Criteria for Warning Signs or Severe Dengue, Regardless of Dengue Serostatus at Baseline, Up to Approximately 3 Years Postvaccination | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA. Clinical evaluation for presence of dengue with warning signs or severe dengue will be conducted by an investigator or medically qualified designee, based on pre-specified criteria.
Percentage of Participants Experiencing Symptomatic (Regardless of Fever) VCD Meeting Criteria for Warning Signs or Severe Dengue, by Dengue Serostatus at Baseline, Up to Approximately 3 Years Postvaccination | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA. Clinical evaluation for presence of dengue with warning signs or severe dengue will be conducted by an investigator or medically qualified designee, based on pre-specified criteria.
Percentage of Participants Experiencing Symptomatic (Regardless of Fever) VCD Meeting Criteria for Warning Signs or Severe Dengue, Regardless of Dengue Serostatus at Baseline, Up to Approximately 5 Years Postvaccination | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA. Clinical evaluation for presence of dengue with warning signs or severe dengue will be conducted by an investigator or medically qualified designee, based on pre-specified criteria.
Percentage of Participants Experiencing Symptomatic (Regardless of Fever) VCD Meeting Criteria for Warning Signs or Severe Dengue, by Dengue Serostatus at Baseline, Up to Approximately 5 Years Postvaccination | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA. Clinical evaluation for presence of dengue with warning signs or severe dengue will be conducted by an investigator or medically qualified designee, based on pre-specified criteria.
Percentage of Participants Experiencing Hospitalization Resulting from Symptomatic (Regardless of Fever) VCD of Any Severity, Regardless of Dengue Serostatus at Baseline, Up to Approximately 3 Years Postvaccination | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Hospitalization Resulting from Symptomatic (Regardless of Fever) VCD of Any Severity, by Dengue Serostatus at Baseline, Up to Approximately 3 Years Postvaccination | Up to approximately 3 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Hospitalization Resulting from Symptomatic (Regardless of Fever) VCD of Any Severity, Regardless of Dengue Serostatus at Baseline, Up to Approximately 5 Years Postvaccination | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Percentage of Participants Experiencing Hospitalization Resulting from Symptomatic (Regardless of Fever) VCD of Any Severity, by Dengue Serostatus at Baseline, Up to Approximately 5 Years Postvaccination | Up to approximately 5 years postvaccination
  Fever is defined as presence of body temperature ≥ 100.4 °F. Dengue status will be confirmed by WT RT-PCR or NS1 ELISA.
Reactogenicity and Immunogenicity Subset: Percentage of Participants who are Seropositive as measured by VRNT, by Dengue Serostatus at Baseline | Up to approximately 28 days postvaccination
  Seropositivity for Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Reactogenicity and Immunogenicity Subset: Percentage of Participants who are Seropositive as measured by VRNT, Regardless of Dengue Serostatus at Baseline | Up to approximately 28 days postvaccination
  Seropositivity for Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Reactogenicity and Immunogenicity Subset: Percentage of Participants who Seroconvert as measured by VRNT, by Dengue Serostatus at Baseline | Up to approximately 28 days postvaccination
  Seroconversion rate for Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Reactogenicity and Immunogenicity Subset: Percentage of Participants who Seroconvert as measured by VRNT, Regardless of Dengue Serostatus at Baseline | Up to approximately 28 days postvaccination
  Seroconversion rate for Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Reactogenicity and Immunogenicity Subset: Dengue Virus-Neutralizing Antibody Titers, as Measured by VRNT, by Dengue Serostatus at Baseline | Up to approximately 28 days postvaccination
  Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Reactogenicity and Immunogenicity Subset: Dengue Virus-Neutralizing Antibody Titers, as Measured by VRNT, Regardless of Dengue Serostatus at Baseline | Up to approximately 28 days postvaccination
  Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Reactogenicity and Immunogenicity Subset: Geometric Mean Fold Rises (GMFRs) in Dengue Virus-Neutralizing Antibody Titers, by Dengue Serostatus at Baseline | Baseline (Day 1) and up to approximately 28 days postvaccination
  GMFRs for Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Reactogenicity and Immunogenicity Subset: GMFRs in Dengue Virus-Neutralizing Antibody Titers, Regardless of Dengue Serostatus at Baseline | Baseline (Day 1) and up to approximately 28 days postvaccination
  GMFRs for Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Long-term Immunogenicity Subset: Percentage of Participants who are Seropositive, as measured by VRNT, by Dengue Serostatus at Baseline | Up to approximately 5 years postvaccination
  Seropositivity for Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Long-term Immunogenicity Subset: Percentage of Participants who are Seropositive, as measured by VRNT, Regardless of Dengue Serostatus at Baseline | Up to approximately 5 years postvaccination
  Seropositivity for Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Long-term Immunogenicity Subset: Percentage of Participants who Seroconvert, as measured by VRNT, by Dengue Serostatus at Baseline | Up to approximately 5 years postvaccination
  Seroconversion rate for Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Long-term Immunogenicity Subset: Percentage of Participants who Seroconvert as measured by VRNT, Regardless of Dengue Serostatus at Baseline | Up to approximately 5 years postvaccination
  Seroconversion rate for Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Long-term Immunogenicity Subset: Dengue Virus-Neutralizing Antibody Titers, as Measured by VRNT, by Dengue Serostatus at Baseline | Up to approximately 5 years postvaccination
  Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.
Long-term Immunogenicity Subset: Dengue Virus-Neutralizing Antibody Titers, as Measured by VRNT, Regardless of Dengue Serostatus at Baseline | Up to approximately 5 years postvaccination
  Dengue virus-neutralizing antibody titers for 4 dengue serotypes (DENV-1, DENV-2, DENV-3, DENV-4) as measured by VRNT will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (29):
- Indonesia (5):
  - Jatinegara Primary Health Center ( Site 0102), East Jakarta, Jakarta Special Capital Region
  - Cipayung Primary Health Center ( Site 0105), East Jakarta, Jakarta Special Capital Region
  - Dr Cipto Mangunkusumo Hospital-Pediatrics ( Site 0101), Jakarta, Jakarta Special Capital Region
  - Kelapa Gading Primary Health Center ( Site 0104), North Jakarta, Jakarta Special Capital Region
  - Pasar Minggu Primary Health Center ( Site 0103), South Jakarta, Jakarta Special Capital Region
- Malaysia (6):
  - University Malaya Medical Centre-Department of Paediatrics ( Site 0025), Lembah Pantai, Kuala Lumpur
  - Hospital Sibu ( Site 0021), Sibu, Sarawak
  - Hospital Ampang ( Site 0028), Ampang, Selangor
  - Hospital Al-Sultan Abdullah - Universiti Teknologi MARA ( Site 0029), Bandar Puncak Alam, Selangor
  - Sunway Medical Centre ( Site 0027), Petaling Jaya, Selangor
  - Hospital Tunku Azizah-Paediatric ( Site 0022), Kuala Lumpur
- Philippines (6):
  - Health Index Multispecialty And Lying-In Clinic ( Site 0042), Bacoor, Cavite
  - Chong Hua Hospital ( Site 0051), Cebu City, Cebu
  - Norzel Medical and Diagnostic Clinic Foundation Corp ( Site 0044), Cebu City, Central Visayas (Region VII)
  - West Visayas State University Medical Center ( Site 0045), Iloilo City, Iloilo
  - Philippine General Hospital ( Site 0041), Manila, National Capital Region
  - University of the Philippines Manila ( Site 0047), Metro Manila, National Capital Region
- Singapore (3):
  - National University Hospital-Paediatrics ( Site 0001), Singapore, Central Singapore
  - KK Women's and Children's Hospital ( Site 0002), Singapore, Central Singapore
  - Tan Tock Seng Hospital ( Site 0003), Singapore, Central Singapore
- Thailand (9):
  - Chulalongkorn University-Pediatrics ( Site 0063), Bangkok, Bangkok
  - Faculty of Tropical Medicine, Mahidol University ( Site 0062), Bangkok, Bangkok
  - Queen Sirikit National Institute of Child Health-Pediatric Infectious Disease ( Site 0071), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital-Pediatric Infectious Diseases ( Site 0065), Bangkok, Bangkok
  - Faculty of Tropical Medicine, Mahidol University - Vaccine Trial Centre ( Site 0067), Ratchathewi, Bangkok
  - Faculty of Medicine - Khon Kaen University-Pediatrics ( Site 0064), Amphoe Mueang, Changwat Khon Kaen
  - Thammasat University Hospital-Department of Pediatrics ( Site 0068), Khong Luang, Changwat Pathum Thani
  - Songklanagarind hospital-Department of Pediatrics ( Site 0061), Hat Yai, Changwat Songkhla
  - Maharaj Nakorn Chiang Mai Hospital ( Site 0066), Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com